CLINICAL TRIAL: NCT00135369
Title: A Phase 3 Study Switching HIV-1 Infected Subjects With an Undetectable Viral Load From a HAART Regimen Dosed Twice Daily or More Frequently to a Once-Daily HAART Regimen
Brief Title: Switching HIV-1 Infected Subjects From a Highly Active Anti-Retroviral Treatment (HAART) Regimen Dosed Twice Daily or More Frequently to a Once-Daily Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI455-135
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: HIV-AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Lamivudine; efavirenz

INTERVENTIONS:
Drug: stavudine extended-release, lamivudine, efavirenz

SUMMARY:
The purpose of this study is to demonstrate that virologically controlled HIV-infected individuals can successfully switch from a standard-of-care regimen dosed twice-daily or more frequently to a simpler once-daily (QD) regimen while maintaining virologic control, as evaluated by the proportion of subjects who continue to have plasma HIV-1 levels <50 copies/mL after switching to a QD regimen.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* 18 years of age or older and weigh at least 40 kg
* Two plasma HIV RNA levels below the limit of quantification (one at least 90 days prior to the screening visit and one within 30 days of the patients baseline visit)
* Currently receiving a standard-of-care HAART regimen with at least one agent being dosed twice-daily or more frequently

Exclusion Criteria:

* Pregnancy, breastfeeding or plans to become pregnant during the study period
* Any prior documented virologic failure to one or more HAART regimens
* Active AIDS-defining opportunistic infection or disease
* Proven or suspected acute hepatitis within 30 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-09; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Efficacy at week 48

SECONDARY OUTCOMES:
Safety, tolerability and efficacy at weeks (wks) 24 and 48; Effect on lipids at wks 24 and 48; Adherence, quality of life changes, treatment satisfaction and preference at wks 12, 24 and 48

CONTACTS AND LOCATIONS:
Locations (47):
- United States (46):
  - Local Institution, Hobson City, Alabama
  - Local Institution, Montgomery, Alabama
  - Local Institution, Phoenix, Arizona
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Los Angeles, California
  - Local Institution, Sacramento, California
  - Local Institution, San Mateo, California
  - Local Institution, Torrance, California
  - Local Institution, Denver, Colorado
  - Local Institution, Norwalk, Connecticut
  - Local Institution, Stratford, Connecticut
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Miami, Florida
  - Local Institution, Miami Beach, Florida
  - Local Institution, Pensacola, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Decatur, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Indianapolis, Indiana
  - Local Institution, New Orleans, Louisiana
  - Local Institution, Baltimore, Maryland
  - Local Institution, Boston, Massachusetts
  - Local Institution, Berkley, Michigan
  - Local Institution, Detroit, Michigan
  - Local Institution, St Louis, Missouri
  - Local Institution, Las Vegas, Nevada
  - Local Institution, Hackensack, New Jersey
  - Local Institution, Jersey City, New Jersey
  - Local Institution, Neptune City, New Jersey
  - Local Institution, Somers Point, New Jersey
  - Local Institution, Manhasset, New York
  - Local Institution, New York, New York
  - Local Institution, The Bronx, New York
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Huntersville, North Carolina
  - Local Institution, Washington, North Carolina
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Reading, Pennsylvania
  - Local Institution, Dallas, Texas
  - Local Institution, Galveston, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Annandale, Virginia
  - Local Institution, Hampton, Virginia
  - Local Institution, Seattle, Washington
- Local Institution, San Juan, Puerto Rico